CLINICAL TRIAL: NCT06886464
Title: The Prevention of Nephrotoxin-Induced Acute Kidney Injury Using Cilastatin (PONTiAK) Trial: A Phase 2B Vanguard Design, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Prevention of Nephrotoxin-Induced Acute Kidney Injury Using Cilastatin
Acronym: PONTiAK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew James (Other)
Collaborators: Alberta Health services (Other); University of Alberta (Other)
Responsible Party: Sponsor-Investigator, Matthew James, Sponsor-Investigator, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NEPH24-1191
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Nephrotoxic; Cilastatin
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cilastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cilastatin Intervention (Experimental): Patients in this Arm will receive the Investigational Medicinal Product- Cilastatin
  Interventions: Drug: Cilastatin Sodium
- Placebo Control (Placebo Comparator): Patients in this Arm will receive placebo
  Interventions: Drug: Placebo-Saline

INTERVENTIONS:
Drug: Cilastatin Sodium — Intravenous cilastatin reconstituted in normal saline solution
  Other Names: Renal dehydropeptidase inhibitor
  Arms: Cilastatin Intervention
Drug: Placebo-Saline — Identical looking normal saline solution
  Other Names: Control
  Arms: Placebo Control

SUMMARY:
The goal of this clinical trial is to repurpose cilastatin for preventing acute kidney injury (AKI) in hospitalized patients receiving nephrotoxic medications. The trial will evaluate the efficacy of the re-purposed drug.

The main questions it aims to answer are:

- whether cilastatin will prevent nephrotoxic AKI in hospitalized patients.

Researchers will compare the drug cilastatin to a placebo (a look-alike substance that contains no drug) to see if drug cilastatin works to prevent AKI in hospitalized patients receiving nephrotoxic medications.

Participants will:

* Receive drug Cilastatin or a placebo intravenously every 6 hours for up to 24 hours after last exposure to nephrotoxic medication
* Have blood test for kidney function every day they are on treatment.
* Have a follow-up blood test at 90 days after randomization
* Have a telephone survey at 90 days after randomization

DETAILED DESCRIPTION:
BACKGROUND People living with chronic diseases frequently require hospitalization, where they are often exposed to a variety of medications. Common medications include drugs for the treatment of cancer, immunosuppression for organ transplantation or autoimmune conditions, antibiotics for infections, and contrast dyes for imaging procedures. Many of these medications can be nephrotoxic and cause iatrogenic acute kidney injury (AKI) in 25% of hospitalized patients, especially among those receiving combinations of multiple medications. The long-term consequences of AKI are many, and include prolonged hospitalization, increased risk of readmission, progression of chronic kidney disease (CKD), and kidney failure. AKI also affects other organ systems and increases the risk of major adverse cardiovascular (CV) events and death. AKI has a profound effect on long-term patient outcomes and places a high burden on the health system by both increasing resource use for acute care as well as those for long-term chronic disease management.

The incidence of AKI has been rising by 10% annually and is highest in people aged 65 and older and among those with pre-existing chronic diseases. As more patients experience AKI, the health burden resulting from these outcomes has become increasingly apparent, with rising rates of progression to CKD, kidney failure, CV events and death. Although nephrotoxic AKI is common and associated with poor outcomes, there is currently a lack of effective preventive strategies other than drug avoidance, which is suboptimal as it denies vulnerable patients from receiving many effective medical therapies.

Clinical Issue and Opportunity:

Nephrotoxic AKI is common among hospitalized patients and there are currently no pharmacologic therapies available for prevention. The Nephrotoxic Injury Negated by Just-In-Time Action (NINJA) research initiative has developed, implemented, and evaluated strategies to identify patients at high risk of nephrotoxic AKI, with the objective of improving identification of high risk patients and reducing harm related to AKI . Several studies employing NINJA criteria have demonstrated an incidence of nephrotoxic AKI of 20-30% among hospitalized patients with multiple medication exposures, including with antibiotics (vancomycin, aminoglycosides), radiographic contrast dye, and calcineurin inhibitors identified among the most commonly associated agents. In hospitalized adults in North America, antibiotics and iodinated contrast are implicated in more than half of all nephrotoxic AKI. Trying to avoid exposure to these medications is suboptimal as it denies patients from receiving the best available therapies. The implementation of a common computerized clinical information system across all hospitals in Alberta provides an opportunity to efficiently identify patients with high risk nephrotoxic medication exposures, and test interventions to prevent AKI and its downstream consequences.

Current Evidence:

CIHR funded studies from our institution and others have identified tubular uptake of nephrotoxins as a major contributor to the pathogenesis of AKI. Dipeptidase-1 (DPEP1) and megalin (LRP2) are proteins that contribute to the uptake of nephrotoxic drugs in the proximal tubules of the kidney. DPEP1 is also a major non-classical leukocyte adhesion receptor that is critical in neutrophil and inflammatory monocyte recruitment to the kidney.

Cilastatin is a small molecule developed and approved for human use as an enzymatic DPEP1 inhibitor to prevent degradation of the antibiotic imipenem. Through the inhibition of DPEP1 and LRP2, cilastatin has proven effective in preventing tubular drug uptake and kidney injury in cell culture and animal models of nephrotoxic AKI from contrast, vancomycin, gentamicin, cisplatin, and cyclosporine. Cilastatin also prevents DPEP1-mediated kidney injury from a variety of causes mediated by inflammation. For these reasons, cilastatin has been indirectly tested in human studies for nephrotoxic AKI prevention, using imipenem-cilastatin formulations approved for clinical use.

A systematic review identified 10 studies (5 RCTs, n=535 patients; 5 observational comparative effectiveness studies n=6,198) that evaluated the nephroprotective effects of imipenem-cilastatin in patients receiving a variety of nephrotoxic medications including calcineurin inhibitors, antibiotics, and chemotherapy. All identified studies reported lower risk of kidney injury (pooled risk ratio 0.54 [95% CI, 0.41 to 0.72] and/or better kidney function between 7 to 30 days after treatment among patients receiving imipenem-cilastatin than comparator groups.

Rationale for Study:

Repurposing cilastatin to target tubular toxin/drug uptake and renal inflammation represents a highly promising and scientifically rational approach to protect the kidney from nephrotoxic AKI and ultimately improve kidney and CV outcomes for patients.

The PONTiAK Study will apply innovative electronic recruitment and data collection methods to complete a randomized Study to efficiently generate new evidence on the efficacy of this treatment strategy. Collectively, the Study will produce valid and generalizable results that will not only inform a pivotal phase 3 Study but also accelerate methods for efficiently and effectively conducting such a clinical Study needed for eventual drug approval. If cilastatin reduces the incidence of nephrotoxin-induced AKI by 10%, it would significantly change clinical practice, preventing more than 10,000 episodes of AKI in Canada each year. This significant AKI reduction has the potential to reduce hospitalization and downstream adverse kidney and CV events, saving ~$78 million annually.

STUDY DESIGN AND WORKFLOW

The PONTiAK Study is a randomized, double blind, placebo-controlled superiority study in hospitalized adults at risk of nephrotoxic AKI. Eligible Participants will be identified using a computer-enabled case finding algorithm for patients with nephrotoxic medication exposures implemented in the common clinical information system called Connect Care used in the six largest hospitals in Alberta. The case finding approach will be adapted from NINJA, an evidence-based algorithm defined by exposure to three medications on the same day from an evidence-based list of 47 drugs from 7 medication classes (plus radiocontrast dyes), or prescription of an aminoglycoside antibiotic or vancomycin for 3 or more days. NINJA is a validated approach to enrich for identification of hospitalized patients at high risk of AKI. Patients meeting the nephrotoxin exposure criteria with an active order for a medication that mediates AKI via DPEP1/LRP2 uptake will be identified daily and approached to obtain informed consent then randomized 1:1 to cilastatin or placebo using a central web-based system. In addition to hospitalized patients, patients receiving eligible chemotherapeutics drugs (eg. platins) in day medicine units of hospitals will also be identified by the algorithm and approached for recruitment.

Treatment with IV cilastatin or matching placebo will be initiated as soon as possible after randomization and continued for up to 24 hours after last exposure to nephrotoxic medication for medications requiring repeated dosing, hospital discharge, or initiation of dialysis. Day Medicine patients will receive IV cilastatin or matching placebo one time immediately before receiving the nephrotoxic medication (typically at the time of pre-medication with IV fluid, anti-emetic, and analgesic administration). The study drug may be discontinued at any time based upon the patient's attending physician's or site investigator's judgement.

Participants will be followed daily in hospital following randomization for the duration of nephrotoxic medication exposure plus 48 hours or until hospital discharge. During this period daily measurements of kidney function (serum creatinine) will be collected in a standardized manner according to the NINJA lab testing algorithm to ascertain the primary outcome of AKI. Participants will also have vital signs and urine output results recorded daily throughout the treatment period and for 48 hours following the end of nephrotoxic medication treatment. Day Medicine patients will have vital signs recorded before and after IMP/placebo infusion, urine output recorded at the end of treatment with cisplatin or carboplatin, and blood work for kidney function done before IMP/placebo infusion and on day 2 and day 7 after nephrotoxic medication administration.

Adverse events will be recorded daily throughout the duration of treatment plus 48 hours. All Participants will also receive follow-up at 30 days following randomization, which will include electronic medical chart review, and assessment by telephone to ascertain the secondary outcomes of the study. To the extent possible, any adverse events that are deemed study drug-related and are ongoing at discharge will be followed-up to resolution or until a determination is made that the unresolved event is stable.

Consent will also be sought from all participants for linkage to routinely collected administrative health data to measure major adverse kidney and cardiovascular outcomes over an extended total of two years follow-up from study enrollment.

SAMPLE SIZE The Study will recruit 698 patients (349 per arm) to achieve 85% power to detect a 10% absolute risk reduction in the incidence of AKI from 25% in the placebo arm to 15% in the cilastatin arm, with a two-sided type 1 error rate of 0.05. The minimal clinically important difference for powering assumptions for the PONTiAK trial are informed by recommendations from existing literature on the design of AKI prevention clinical trials. Ten trials of imipenem-cilastatin versus placebo have been conducted in adults, and our updated systematic review produced a pooled odds ratio for AKI of 0.42 (95% CI 0.26-0.69), with a corresponding absolute risk reduction of 32% (95% CI 16 -77%). The investigators conducted power analysis by simulation considering a substantially smaller minimum clinically important absolute difference in AKI incidence of 10%. Assuming two event probabilities of 0.25 (placebo) and 0.15 (cilastatin) drawn from a binomial distribution, a two-sided type 1 error rate of 0.05 (applying a chi-square test), using at least 10,000 replicates of the experiment, the investigators found that 349 participants per arm would confer a power of 85% to the PONTiAK trial. With this sample size the trial will still have a power of 80% even with up to a 10% loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Active treatment with an eligible nephrotoxic medication- IV vancomycin, IV aminoglycoside (gentamicin or tobramycin), IV calcineurin inhibitor (cyclosporine or tacrolimus), or IV or intraperitoneal platin-based chemotherapy or ifosfamide; or intraarterial radiographic contrast with two or more high-risk nephrotoxic medication exposures according to the NINJA algorithm.
* Able to provide informed consent or have an authorized representative available and willing to give written informed consent after being properly informed of the nature and risks of the Study.

Exclusion Criteria:

* Stage 3 AKI based on Kidney Disease Improving Global Outcomes (KDIGO) SCr or urine output criteria, or receipt of short-term dialysis.
* Category G5 CKD (defined as a CKD-EPI eGFR or <15 mL/min/1.73 m2) or being treated with maintenance dialysis or a kidney transplant.
* Pregnancy or lactation
* Known hypersensitivity to imipenem-cilastatin.
* Active or recent treatment (within 48 hours) with imipenem-cilastatin
* Active or recent treatment (within 48 hours) with probenecid (medication used for gout prevention that inhibits cilastatin excretion and decreases plasma clearance)
* Treatment with another investigational medicinal product or participation in another interventional Study within 30 days
* Inability to comply with the requirements of the Study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants developing AKI | 7 days after administration of a nephrotoxic medication
  Evaluation of Acute Kidney Injury (AKI) according to KDIGO serum creatinine (SCr) criteria; ≥ 26 mmol/L (0.3 mg/dL) increase in SCr within 48 hours or ≥50% increase in SCr within 7 days

SECONDARY OUTCOMES:
Number of participants developing stage-1, stage-2, and stage-3 AKI | Within 30 days of administration of nephrotoxic medication
  * Stage 1; SCr increase ≥26 μmol/L (≥0.3 mg/dL) or 1.5 - 1.9 times baseline.
  * Stage 2; SCr increase 2.0 - 2.9 times baseline.
  * Stage 3; SCr increase ≥3.0 times baseline OR increase in SCr ≥353.6 μmol/L (≥4.0 mg/dL) OR initiation of dialysis
Number of participants needing dialysis | Within 30 days of administration of nephrotoxic medication
  Receipt of short or long-term dialysis
Number of days admitted to hospital | Within 30 days of receiving nephrotoxic medication
  Hospital length of stay
Measurement of eGFR and Cystatin C | 90 days from study enrollment.
  Kidney function based on SCr (eGFRSCr) and Cystatin C (eGFRCysC).
Number of participants with SCr 1.5 times less than baseline | 90 days from study enrollment.
  Persistent decrease in kidney function, defined by SCr > 26 μmol/L (≥0.3 mg/dL) or 1.5 times baseline
Measurement of urinary albumin to creatinine ratio (ACR) | 90 days from study enrollment.
  Kidney damage based on urinary albumin to creatinine ratio (ACR)
Hospital readmission | 90 days from study enrollment.
  Readmission to a hospital following a discharge (does not include interfacility transfer)
All-cause mortality | 90 days from study enrollment.
  Death from any cause
Physical and mental functional | 90 days from study enrollment.
  Physical and mental functional status based on short-form-12 (SF-12)

OTHER OUTCOMES:
Number of participants developing Major Adverse Kidney Event (MAKE) | 2 years from study enrollment
  Major adverse kidney (maintenance KRT, 40% decline in eGFRSCr, or death) event (MAKE) determined via administrative data linkage.
Major Adverse Cardiovascular Endpoint (MACE) | 2 years from study enrollment
  Major adverse cardiovascular (myocardial infarction, stroke, hospitalization for heart failure or death) event (MACE) determined from patient administrative data.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T James, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliott MJ, Fiest KM, Love S, Birdsell D, Loth M, Dumka H, Rana B, Shommu N, Benterud E, Gil S, Acharya D, Harrison TG, Pannu N, James MT. Patient Preferences and Priorities for the Design of an Acute Kidney Injury Prevention Trial: Findings from a Consensus Workshop. Kidney360. 2024 Oct 1;5(10):1455-1465. doi: 10.34067/KID.0000000000000554. Epub 2024 Aug 15. PMID 39146029
- [Background] Acharya D, Ghanim F, Harrison TG, Scory TD, Shommu N, Ronksley PE, Elliott MJ, Collister D, Pannu N, James MT. Nephroprotective Effects of Cilastatin in People at Risk of Acute Kidney Injury: A Systematic Review and Meta-analysis. Kidney Med. 2024 Oct 11;6(12):100913. doi: 10.1016/j.xkme.2024.100913. eCollection 2024 Dec. PMID 39583177
- See also: Alberta Health Services Connect Care. — https://www.albertahealthservices.ca/cis/cis.aspx